CLINICAL TRIAL: NCT00745602
Title: The Effect of Atrial Fibrillation Hemodynamics on Regulation of Cerebral Blood Flow
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Could not get funding
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: UTSW IRB 092007-020
Record Dates: First submitted 2008-08-29; First posted 2008-09-03 (Estimated); Last update posted 2019-01-09 (Actual); Status verified 2019-01

CONDITIONS: Atrial Fibrillation
Keywords: direct current cardioversion, cerebral blood flow
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): Patients referred for elective direct current cardioversion (DCCV) of atrial fibrillation.
  Interventions: Procedure: non-invasive testing

INTERVENTIONS:
Procedure: non-invasive testing — non-invasive tests including Transcranial Doppler ultrasound (TCD), manual cuff blood pressure (BP), beat to beat BP monitoring by a Portapress monitor, and respiratory tidal CO2

SUMMARY:
The proposed research will investigate whether the irregular effects of atrial fibrillation on the body's circulation directly impacts the regulation of cerebral blood flow. To further delineate this finding, investigation of these potential effects will include differences in postural positioning. This data will be used to further understand the overall hemodynamic effects of atrial fibrillation on extra-cardiac organs of the body.

DETAILED DESCRIPTION:
This is a prospective study evaluating 10 subjects referred for elective direct current cardioversion (DCCV) of atrial fibrillation. Subjects will be seen at Parkland Health and Hospital System.

After full consent is obtained and explanation of the research, each subject will undergo a series of entirely non-invasive tests including Transcranial Doppler ultrasound (TCD), manual cuff blood pressure (BP), beat to beat BP monitoring by a Portapress monitor, and respiratory tidal CO2. These measurements will be taken after laying the patient in a supine position for 10 minutes and subsequently after standing for 10 minutes. Measurements will also be taken after full body squat -stand repetition at 20 second intervals (0.05 Hz) x 5 minutes. Patients who are unable to squat may rise from a seated position on a chair. This protocol has been easy to follow even for debilitated patients with Alzheimers Disease in Dr. Zhang and Dr. Levine's laboratory. The subject will then undergo elective DCCV as planned for standard of care. The above measurements and with respective body positions will then be repeated 30 minutes later if the patient has been successfully converted to normal sinus rhythm by DCCV.

The experimental testing will take approximately 1 ½ to 2 hours to complete.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with atrial fibrillation scheduled for DCCV
* Subjects must be at least 18 years of age
* Subjects must have the ability to understand and sign informed consent and be willing to comply with full testing and evaluation

Exclusion Criteria:

* Subjects in sinus rhythm without assessment of any prior atrial fibrillation by this research team
* Subjects unable to understand and given informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2007-10; Primary Completion 2009-10 (Estimated); Study Completion 2009-10 (Estimated)

PRIMARY OUTCOMES:
to determine whether the irregular effects of atrial fibrillation on the body's circulation directly impacts the regulation of cerebral blood flow | 0

CONTACTS AND LOCATIONS:
Overall Officials: Jose A Joglar, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- UT Southwestern Medical Center, Dallas, Texas, United States